CLINICAL TRIAL: NCT06129825
Title: Pharmacologic Induction of Tolerance for Hypoxia & Hypothermia
Acronym: PhITHy-Ho
Status: Active, not recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Allan Doctor, MD, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00108068
Record Dates: First submitted 2023-10-18; First posted 2023-11-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypothermia; Hypoxia; Mountain Sickness
MeSH Terms: conditions — Hypothermia; Hypoxia; Altitude Sickness | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh human blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteers: Healthy Adults Volunteers >/= 18yrs of age without acute or chronic illness.
  Interventions: Other: Prospective

INTERVENTIONS:
Other: Prospective — Single arm, healthy adult volunteers for blood donation.

SUMMARY:
Warfighter Performance Optimization in Extreme Environments remains an area of important and intense investigation, with the following goals: (1) Optimize, sustain and augment medical readiness and physiological/ psychological performance in extreme and hazardous military operational environments and (2) develop joint DoD countermeasures and guidance to sustain performance, assess physiological status, and reduce injury risk in extreme and hazardous operational environments. Successful and safe outcomes in extreme and hazardous operational environments require that warfighters maintain optimum cognitive and exercise performance during physiologic stress. Extreme environmental conditions encountered in such environments include warfighter exposure to hypoxia and hypothermia, alone or in combination. Both hypoxia and hypothermia undermine O2 delivery system homeostasis, imposing dangerous constraints upon warfighter cognitive and exercise capacity.

While red blood cells (RBCs) are commonly recognized as O2 transport agents, their function as a key signaling and control node in O2 system delivery homeostasis is newly appreciated. Through O2 content-responsive modulation of RBC energetics, biomechanics, O2 affinity and control of vasoactive effectors in plasma - RBCs coordinate stabilizing responses of the lung, heart, vascular tree and autonomic nervous system - in a fashion that maintains O2 delivery system homeostasis in the setting of either reduced O2 availability (hypobaric hypoxia) or increased O2 demand (hypothermia). Human RBCs demonstrate adaptive responses to exercise, hypoxia and hypothermia - these changes are commonly appreciated as a key element enabling high altitude adaptation. However, under conditions of hypoxia and hypothermia, without prior adaptation, RBC performance is adversely impacted and limits the dynamic range of stress adaptation for O2 delivery homeostasis - therefore limiting warfighter exercise capacity and cognitive performance in extreme environments, such as during acute mountain sickness.

DETAILED DESCRIPTION:
The investigator's strategy is to: (a) repurpose approved drugs with potential for salutary effect upon RBC performance attributes that contribute to O2 delivery homeostasis during stress and (b) efficiently identify lead candidates through sequential evaluation in relevant and rigorous benchtop and in vivo models that include examination for gender-specific effects. Our assay platforms are selected to characterize RBC physiology relevant to O2 delivery, with focus upon RBC O2 affinity, energetics, biomechanics, vascular interaction and control of regional blood flow. The investigator will sample RBC suspensions serially (0, 1,3h) and quantify the RBC performance attributes across the range of modeled environmental extremes, defining RBC performance constraint as > 20% impairment in each attribute and determine pharmacologic rescue (defined as > 20% improvement in each attribute) using mixed model RM-ANOVA, as a function of gender. The investigator will power analysis to 80% at a<5%; based on our published data with these assays and experience, this requires 10-15 subjects/group. Drug candidates with evidence of PhIT-HyHo potential will advance to in vivo screening, prioritized by the number of RBC attributes rescued per drug. Specific description of our approach to evaluate each RBC performance attribute follows.

RBC performance attributes will be quantified under controlled conditions (Temperature: 28 - 37°C; pO2: 50 - 100 Torr, alone and in combination in our temperature-controlled thin film tonometer38 (NB temperature simulates hypothermic body temperature): (a) glycolytic flux, (b) resilience to oxidative stress, (c) deformability & aggregation, (d) O2 affinity and Bohr effect, (e) vasoactivity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >/= 18years of age.
* Subject weighs a minimum of 110lbs
* Subject must be generally healthy individual

Exclusion Criteria:

* Suspected or diagnosed with ongoing (chronic) or acute infection
* Pregnant
* Non-English speaking
* Ages 89 and over

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adults 18-88 years of age.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Drug candidate effects on RBC energy metabolism | 18-24months
  The Investigator will specifically focus on relative glycolytic and pentose phosphate pathway flux, to determine robustness of RBC antioxidant capacity. Flux analysis will be performed by metabolomics (mass spectrometry).

SECONDARY OUTCOMES:
Drug candidate effects on RBC resilience to oxidative stress. | 18-24months
  The Investigator will assess robustness of RBC antioxidant systems following in vitro incubation in an oxidative environment. Outcome measures will include the ability of RBC's to scavenge oxidants including superoxide and hydrogen peroxide, RBC lysis and oxidative changes in RBC membrane proteins.

OTHER OUTCOMES:
Drug candidate effects on RBC deformability and aggregation. | 18-24months
  RBC deformability will be assessed by ektacytometry and Brillouin microscopy. Measurements will include elongation index (ability of RBC's to elongate as a function of shear) in addition to a non-shear assessment of RBC deformability. Aggregation will be assessed by syllectometry.
Drug candidate effects on RBC 02 affinity and Bohr effect. | 18-24months
  This will be assessed using the HEMOX analyzer and thin film tonometry (with gas mix blending) to determine hemoglobin p50 shift (i.e., the partial pressure of oxygen at which hemoglobin is 50% saturated with oxygen) and the ability of hemoglobin O2 affinity to respond to pH.
Drug candidate effects on RBC 02 vasoactivity. | 18-24months
  RBC's will be tested in a bio-assay containing aortic tissue to determine their dilatory capacity under hypoxia and their constriction properties under normoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Doctor, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided